CLINICAL TRIAL: NCT01912898
Title: Development of Non-invasive Method for Quantifying Vitamin D Levels in the Body Using Spectroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0009-13
Record Dates: First submitted 2013-07-17; First posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-02

CONDITIONS: Deficiency of Vitamin D Blood Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1
  Interventions: Device: No intervention,The group with vitamin D deficient will be treated by the Endocrinology Department by loading of vitamin D

INTERVENTIONS:
Device: No intervention,The group with vitamin D deficient will be treated by the Endocrinology Department by loading of vitamin D

SUMMARY:
Lack in vitamin D reduces the absorption of calcium in the body; accelerates bone loss tnd may increase the risk of fractures due to osteoporosis. An algorithm that will allow immadiate and non -invasiv quanification of vitamin D levels will shorten the time of diagnosis; reduce lab costs and prevent hazards or discomfort to patient associated with a blood test.

The goal of the study is therfore to develop a non invasive method for quanitifying vitamin D levels in the body using specroscopy.

40 subgects will be recruited: 20 hospitalized patients in the endocrinology departmet, diagnosed with vitamin D deficiency. and 20 healthy subjects. Spectroscopy will be used with wisible lighy on the subject's skin and middle infrared (MIR) on the blood sample to find correlation with the chemical lab test results.

DETAILED DESCRIPTION:
Lack in vitamin D reduces the absorvtion of calcium in the body, accelerates bone loss and may increase the risk of fractures due to osteoporosis. Vitamin D can be ingested by foods and specific supplements, but the main source for the vitamin is synthesis in the skin by usin sun radiation. Today, quanitification of vitamin D levels is performed using a blood test. Mostly; the physician will send the patient to check the levels and vitamin D if he suffers from osteoporosis, renal inpairment, suspected for activity of the thyroid gland; tubeculosis or sacoidosis.

studies have shown that it is possible to quantify the different elements in the contents of the blood, such as melanin and hemoglobin, using spectroscopy of the skin (Zonion et al, 2001; Tseng et al, 2009), but to the investigators knowledge, the identification of levels and vitamin D in similar means has not been reported in professional literature.

The rationale for this research: an algorithm that will allow immediate and non- invasive quantification of vitamin D levels will shorten the time of diagnosis, reduce lab costs and prevent hazards or dicomfort to the patientassociated with a blood test.

Methods:

40 subjects aged 18-65 will be recruted for this research: 20 patients be recruited from the population of patients in the endocrinology department who were diagnosed withe osteoporosis. Also, 20 healthy subjects will be recruited.

All participants will be able to understand the study protcol and sign a consent form independetly.

In this study, the investigators will look for a correlation between the results of conventional blood test for detection of vitamin D levels in the blood and the results of measurements of spectral examinations that will be performed on various locations on the upper body of the subject. These measurements will take place in Hillel Yaffe Medical Center as the subject arrives to the Endocrinolgy department for the blood test. Visible lighy spectrometer (manufactured by Ocean Optics, USB 2000 model), connected to a optical fiber (manufactured by Ocean Optics, diameter 1 mm) will be used. The measurement will use a light soure (Fiberoptics Technology lnc. company. Model SOL-R150)Connected also to an optical fiber. Both ends of the fiber will be positioned on the upper body of the patient one of two configurations: for areas withe greater thickness, e.g. the forearm, the fibers would be placed next to each other on the same side of the limb to measure the return of the light, and in areas with smaller tissue thickness, e.g. finger tip, the fibers will be placed to bothe sides of an organ and record light transmission through the target.

First' the investigators will attempt to find correlation between the spectral analysis results of the visible wavelengths and the blood test. Then the investigators will further compare the subjects blood sampled usind FTIR spectrometer in the mid infrared (device manufactured by Oriel, Model MIR8025). The device is equpped with plug-ATR (Attenuated Total Reflectance) and allows testing of a small sample of fluids. Vials of samples delivered to Rupin on foil-wrapped test using a cooler with ice will be tested in Ruppin on the day of extraction. The samples will be disposed of as biological waste.

Trial protocol:

Each subject will arriv at the Endocrinology department in Hillel Yaffe Medical Center. The subject will rea and sign an informed consent form for pariticipation in the study. The subject will fill out a short questionnaire reporting on the nature of sun exposure, dietary habits and chronic medications.

then the testw will be perfomed:

1. blood test for vitamin D 25 level. Accprdomg to the results we defined the grups. test results with values of equal to or above 30ng/ml is Regultory Group
2. blood test results of vitamin D25 less than 20mg/ml the subgect will accepted loading of vitamin D3 dose of 75,000 IU. and will be follow up dynamiclly increase the level of vitamin D in the blood. The blood test will be taken in time ziro, after four hours , 24 hours and 48 hours after taking the drug.
3. Blood test for vitamin D level 25 (serum) in emty tube protected from ligh,will be taken to Roppin for spectral test.
4. Test using the spectrometer: two fiber optic guided by the researchers on different places on the torso of the patient, when one side of the fiber optic is connected to a light source and the anther optical fiber end is connected to the spectrometer.

There is no expected risk or discomfort to the subject beyound the risk associated with regular blood tests. Spectral test to be held Ruppin on the patient's blood samples, as described in the methods, and will not require the presence of the patient.

Data analysis:

Several algorithms will be developed to be used on the spectral database, in order to identify individuals suffering from vitamin D dificuency.

The data processing will be as follows:

1. Statistical analyzes will be carried out using regression methods to find correlation between the level of vitamin D quantified with laboratory chmical test of the blood and spectral measurements in the visible light as performed at the hospital in different areas of the body.
2. Statistical analyzes will be carried out using regression methods to find correlation between the level of vitamin D quantified with lboratory chemical test of the blood ans spectral measurements in middle infraed (MIR), as preformed on blood samples taken from subjects.
3. The tested population will be divided into two groups according to the blood test results: subjects defined as having vitamin D dificiency and subjects classified as having normal vitamin D levels. Clustering methods of analysis will be carried out, such as PCA and LDA,to find distinguishing characteristic between the two populations.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Ages between 18 - 120

Exclusion Criteria:

* pregnant
* cannot understand or sign a consent form independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 subjects aged 18-65 will be recruted for this research: 20 patients be recruited from the population of patients in the endocrinology department who were diagnosed withe osteoporosis. Also, 20 healthy subjects will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
vitamin D levels | At beseline

CONTACTS AND LOCATIONS:
Overall Officials: Ayelet Tzor, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel